CLINICAL TRIAL: NCT05378685
Title: The Effect of Oral Versus Nasal Intubation on Feeding Outcomes in Neonates Requiring Cardiac Surgery
Brief Title: Nasal vs. Oral Intubation for Neonates Requiring Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Melissa Yildirim, MD, Resident, Pediatrics, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20789
Record Dates: First submitted 2022-05-06; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Congenital Heart Disease; Oral Aversion
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Intubation, Intratracheal

STUDY DESIGN:
Intervention Model Description: Using a random number generator, infants are randomized to oral or nasal intubation by a pediatric cardiac anesthesiologist at the time of surgery. The anesthesiologist may elect to diverge from the randomization based on their clinical judgement and patient safety. Infants are analyzed as treated.
Masking Description: The intubation route (oral or nasal) is obvious and visible to everyone who interacts with the infant postoperatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral (Active Comparator): Infants in this group are endotracheally intubated through their mouth.
  Interventions: Procedure: Endotracheal intubation
- Nasal (Active Comparator): Infants in this group are endotracheally intubated through their nose.
  Interventions: Procedure: Endotracheal intubation

INTERVENTIONS:
Procedure: Endotracheal intubation — The patient is intubated using a laryngoscope and cuffed endotracheal tube. The selection and size of the equipment is at the discretion of the pediatric cardiac anesthesiologist.

SUMMARY:
Often, infants struggle to feed orally after surgery for congenital heart disease and may require supplemental feeding interventions at discharge. In this study, the investigators prospectively randomize infants to oral or nasal endotracheal intubation for surgery and assess postoperative feeding success.

DETAILED DESCRIPTION:
Patients who require cardiac surgery in the neonatal period frequently encounter difficulties reaching full volume oral feeds. These difficulties are related to developmental features, perioperative events, and post-operative oral aversion symptoms. Patients who struggle with oral feeding require longer hospitalizations and frequently require invasive devices for stable nutrition at discharge. The investigators hypothesize that nasal intubation for neonatal cardiac surgery may reduce time to full oral feeds and decrease the proportion of patients requiring discharge feeding tubes.

This is a single-center, prospective randomized control trial of patients less than 2 weeks of age who undergo endotracheal intubation at the time of cardiac surgery. The investigators exclude patients who were <37 weeks corrected gestational age (GA) at surgery, had orofacial or gastrointestinal anomalies, required >5 days of intubation before surgery, or required ECMO or >5 minutes of CPR at any time during the hospitalization. Patients are randomized to nasal (NI) or oral intubation (OI) by a trained pediatric cardiac anesthesiologist at the time of their surgery.

Infants are followed post-operatively until the time of discharge and otherwise receive routine care in the intensive care unit and acute cardiology service. Information regarding feeding milestones is obtained from the electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

* Infants who require surgery for congenital heart disease before 2 weeks of age

Exclusion Criteria:

* < 37 weeks estimated gestational age at the time of surgery
* Orofacial or gastrointestinal anomalies
* Devastating neurologic injury or malformation
* Intubation > 5 days prior to surgery
* > 5 minutes of CPR or ECMO at any time

Max Age: 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Feeding method at discharge | Approximately 1 month after surgery
  Infants are discharged home either fed completely by mouth, fed by nasogastric tube (plus/minus some oral feeds), or gastrostomy tube (plus/minus some oral feeds).

SECONDARY OUTCOMES:
Time to full feeds | Approximately 1 month after surgery
  Infants are assessed for the time to progress to the following feeding milestones: speech pathologist assessment, speech pathologist clearance, NG tube removal, discharge home.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Yildirim, MD, Principal Investigator — UVA Pediatric Intensive Care Unit
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Averin K, Uzark K, Beekman RH 3rd, Willging JP, Pratt J, Manning PB. Postoperative assessment of laryngopharyngeal dysfunction in neonates after Norwood operation. Ann Thorac Surg. 2012 Oct;94(4):1257-61. doi: 10.1016/j.athoracsur.2012.01.009. Epub 2012 Mar 14. PMID 22421593
- [Background] Hehir DA, Easley RB, Byrnes J. Noncardiac Challenges in the Cardiac ICU: Feeding, Growth and Gastrointestinal Complications, Anticoagulation, and Analgesia. World J Pediatr Congenit Heart Surg. 2016 Mar;7(2):199-209. doi: 10.1177/2150135115615847. PMID 26957404
- [Background] Kogon BE, Ramaswamy V, Todd K, Plattner C, Kirshbom PM, Kanter KR, Simsic J. Feeding difficulty in newborns following congenital heart surgery. Congenit Heart Dis. 2007 Sep-Oct;2(5):332-7. doi: 10.1111/j.1747-0803.2007.00121.x. PMID 18377449
- [Background] Piggott KD, Babb J, Yong S, Fakioglu H, Blanco C, DeCampli W, Pourmoghadam K. Risk Factors for Gastrostomy Tube Placement in Single Ventricle Patients Following The Norwood Procedure. Semin Thorac Cardiovasc Surg. 2018 Winter;30(4):443-447. doi: 10.1053/j.semtcvs.2018.02.012. Epub 2018 Feb 9. PMID 29432890
- [Background] Pinelli J, Symington A. Non-nutritive sucking for promoting physiologic stability and nutrition in preterm infants. Cochrane Database Syst Rev. 2005 Oct 19;(4):CD001071. doi: 10.1002/14651858.CD001071.pub2. PMID 16235279
- [Background] Scahill CJ, Graham EM, Atz AM, Bradley SM, Kavarana MN, Zyblewski SC. Preoperative Feeding Neonates With Cardiac Disease. World J Pediatr Congenit Heart Surg. 2017 Jan;8(1):62-68. doi: 10.1177/2150135116668833. PMID 28033074
- [Background] Skinner ML, Halstead LA, Rubinstein CS, Atz AM, Andrews D, Bradley SM. Laryngopharyngeal dysfunction after the Norwood procedure. J Thorac Cardiovasc Surg. 2005 Nov;130(5):1293-301. doi: 10.1016/j.jtcvs.2005.07.013. Epub 2005 Oct 13. PMID 16256781
- [Background] Spence K, Barr P. Nasal versus oral intubation for mechanical ventilation of newborn infants. Cochrane Database Syst Rev. 2000;1999(2):CD000948. doi: 10.1002/14651858.CD000948. PMID 10796391
- [Background] Xue FS, Liao X, Liu KP, Liu Y, Xu YC, Yang QY, Li P, Li CW, Sun HT. The circulatory responses to tracheal intubation in children: a comparison of the oral and nasal routes. Anaesthesia. 2007 Mar;62(3):220-6. doi: 10.1111/j.1365-2044.2007.04939.x. PMID 17300297
- [Derived] Yildirim MI, Spaeder MC, Castro BA, Chamberlain R, Fuzy L, Howard S, McNaull P, Raphael J, Sharma R, Vizzini S, Wielar A, Frank DU. The Impact of Nasal Intubation on Feeding Outcomes in Neonates Requiring Cardiac Surgery: A Randomized Control Trial. Pediatr Cardiol. 2024 Feb;45(2):426-432. doi: 10.1007/s00246-023-03322-7. Epub 2023 Oct 18. PMID 37853163

DOCUMENTS (2):
  • Study Protocol (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT05378685/Prot_000.pdf
  • Informed Consent Form (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/85/NCT05378685/ICF_001.pdf